CLINICAL TRIAL: NCT06028672
Title: Efficacy and Safety of Actinomycin-D With or Without Toripalimab as Fist-Line Treatment in Patients With Gestational Trophoblastic Neoplasia With FIGO Score 5-6: A Multicenter, Open-label, Randomized Controlled Trial
Brief Title: Toripalimab Plus Actinomycin-D as Fist-Line Treatment for GTN With FIGO Score 5-6
Acronym: TA56
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Obstetrics & Gynecology Hospital of Fudan University (Other); Shengjing Hospital (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Henan Cancer Hospital (Other Government); Gansu Provincial Maternal and Child Health Care Hospital (Other); Dalian Maternity and Child Care Hospital (Other); The First Affiliated Hospital of Xiamen University (Other); Sichuan Cancer Hospital and Research Institute (Other); Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Principal Investigator, xiang yang, Professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TA56-GTN-001
Record Dates: First submitted 2023-08-27; First posted 2023-09-08 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Gestational Trophoblastic Neoplasia
Keywords: Gestational Trophoblastic Neoplasia; International Federation of Gynecology and Obstetrics; Toripalimab; Actinomycin-D; Efficacy; Safety
MeSH Terms: conditions — Gestational Trophoblastic Disease | interventions — toripalimab; Dactinomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Toripalimab Plus Actinomycin-D (Experimental): Toripalimab 200mg intravenously(IV) every 2 weeks (Q2W) Actinomycin-D 1.25mg/m2，2mg max dos, intravenously(IV) every 2 weeks (Q2W)
  Interventions: Drug: Toripalimab; Drug: Actinomycin-D
- Actinomycin-D Alone (Active Comparator): Actinomycin-D 1.25mg/m2，2mg max dos, intravenously(IV) every 2 weeks (Q2W)
  Interventions: Drug: Actinomycin-D

INTERVENTIONS:
Drug: Toripalimab — 200mg q2w intravenous
  Arms: Toripalimab Plus Actinomycin-D
Drug: Actinomycin-D — 1.25mg/m2，2mg max dose, q2w, intravenous

SUMMARY:
Whether toripalimab plus actinomycin-D as fist-line treatment can achieve a higher complete response rate than actinomycin-D alone.

Whether an equally high cure rate can be achieved by multi-drug chemotherapy as second-line treatment in patients who have failed fist-line treatment with toripalimab plus actinomycin-D.

Participants will be allocated into two groups. Those in experimental group will receive toripalimab plus actinomycin-D, while those in control group will receive actinomycin-D alone. Treatment will be continued until disease progression, unacceptable toxicity, or withdrawal of consent. Treatment will be completed after 3 consolidation cycles.

DETAILED DESCRIPTION:
The goal of this clinical trial is to evaluate the efficacy and safety of actinomycin-D with or without toripalimab as fist-line treatment in patients with gestational trophoblastic neoplasia with FIGO score 5-6.

Eligible Participants will be randomized into two groups. Those in experimental group will receive toripalimab (200mg q2w intravenous) plus actinomycin-D (1.25mg/m2，2mg max dose, intravenous). While those in control group will receive actinomycin-D (1.25mg/m2，2mg max dose, intravenous) alone. After normalization of serum β-human chorionic gonadotropin (β-hCG) levels, patients will receive 3 cycles of consolidation treatment. Treatment will be continued until completion of treatment, disease progression, unacceptable toxicity, or withdrawal of consent. The primary endpoint is complete remission rate (the proportion of patients achieving complete remission). Secondary endpoints include objective response rate (the proportion of patients achieving complete remission and partial remission), progression-free survival (time from the treatment initiation to disease progression or death, whichever comes first), disease control rate, duration of response, overall survival (time from the treatment initiation to the date of death or last follow-up), duration of response (time from the first evidence of response to disease progression or death, whichever comes first) safety, biomarker, ovarian function and quality of life.

ELIGIBILITY:
Inclusion Criteria:

Diagnosed as GTN: There is a histologic diagnosis of choriocarcinoma or invasive mole. Postmolar GTN: The plateau of β-hCG (±10%) lasts for four measurements over a period of 3 weeks or longer (days 1, 7, 14, 21). There is a rise (>10%) in β-hCG for three consecutive weekly measurements over at least a period of 2 weeks or more (days 1, 7, 14). GTN after nonmolar pregnancy: There is a rise after decease, or a plateau of β-hCG 4 weeks after abortion, ectopic pregnancy, or term delivery. Pregnancy residue or new pregnancy have been ruled out.

Patients with a FIGO score of 5-6. Signed informed consent. No previous immunotherapy, chemotherapy, or radiotherapy. Woman aged 18-60 years. Expected survival ≥ 6 months. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 within 7 days before first dose.

The function of vital organs meets the following requirements: hemoglobin ≥90 g/L, absolute neutrophil count ≥1·5×109/L, platelets ≥100×109/L; creatinine ≤1·5 × upper limit of normal (ULN), urea nitrogen ≤2·5×ULN; total bilirubin ≤1.5×ULN, alanine aminotransferase and aspartate aminotransferase ≤2·5×ULN, INR, PT or APTT ≤1.5×ULN, thyroid stimulating hormone ≤ULN (if thyroid stimulating hormone is abnormal, normal T3 and T4 can also be acceptable).

Exclusion Criteria:

Histologically confirmed placental-site trophoblastic tumor (PSTT) or epithelioid trophoblastic tumor (ETT).

Histologically confirmed primary choriocarcinoma. Other malignancies in the past 3 years. Prior systemic anti-cancer treatment, including chemotherapy and radiotherapy. Live vaccines injected within 30 days before the first dose of study drug; Systemic immune stimulant agent (such as a bacterial or viral vaccine, colony-stimulating factors, interferon, interleukin, and combined vaccine) was used 6 weeks before administration or within the 5 half-lives of the drug, whichever is shorter.

Previous treatment with immunotherapy drugs (including antibodies targeting PD-1, PD-L1, PD-L2, cytotoxic T-lymphocyte-associated protein 4, T-cell receptor, chimeric antigen receptor T-cell therapy, and other immunotherapy).

Known hypersensitivity or allergy to actinomycin-D, toripalimab or any of their excipients.

Any active autoimmune disease requiring systemic treatment during the past 2 years.

History or current status of non-infectious pneumonia requiring steroid treatment.

Receiving steroid hormones (prednisone dose > 10mg/ day) or other immunosuppressants within 14 days before enrollment, excluding those on hormone replacement therapy.

Active infection that requires systemic treatment. Human immunodeficiency virus infection or known acquired immunodeficiency syndrome, active hepatitis B, hepatitis C.

History of psychotropic drug abuse and are unable to withdraw the psychotropic drug, or have mental disorders.

Grade II or higher myocardial ischemia, myocardial infarction or poorly controlled arrhythmia (females with QTc interval ≥470 ms); grade III to IV cardiac insufficiency according to New York Heart Association (NYHA) criteria, or cardiac color Doppler ultrasound evidence of left ventricular ejection fraction <50%; myocardial infarction, NYHA grade II or above heart failure, uncontrolled angina, uncontrolled severe ventricular arrhythmia, clinically significant pericardial disease, or electrocardiogram suggesting acute ischemia or abnormal active conduction system occurring within 6 months before enrolment.

Uncontrollable hypertension (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg, despite with the optimal drug therapy).

Abnormal coagulation (international normalized ratio >1·5×ULN or prothrombin time >ULN+4 seconds or activated partial thromboplastin time >1·5×ULN), with bleeding tendency or undergoing thrombolysis or anticoagulant therapy.

History of cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism within 3 months before enrolment.

Obvious factors affecting oral drug absorption, such as inability to swallow, chronic diarrhea and intestinal obstruction, or sinus or perforation of empty organs within 6 months.

A history of allogeneic stem cell transplantation or organ transplantation. Other reasons as judged by the investigator.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-09-12 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Complete remission rate | up to one year
  The proportion of patients achieving complete remission. Complete remission is defined as normal serum β-hCG level measured for 4 consecutive weeks.

SECONDARY OUTCOMES:
Objective response rate | up to one year
  The proportion of patients with complete or partial response according to serum β-hCG level.
Progression-free survival | up to one year
  The time from the treatment initiation to disease progression or death, whichever comes first. Disease progression is defined as any increase in serum β-hCG level from baseline after 2 cycles of treatment or the presence of new metastatic lesions.
Disease control rate | up to one year
  The proportion of patients with complete response, partial response, or stable disease according to serum β-hCG level.
Duration of response | up to one year
  The time from the first evidence of response to disease progression or death, whichever comes first.
Overall survival | up to one year
  The time from the treatment initiation to the date of death or last follow-up.
Treatment-Emergent Adverse Events [Safety and Tolerability] | up to one year
  Determine frequency and severity of adverse events as assessed by NCI CTCAE (Version 5.0) .
Ovarian function | up to one year
  Ovarian function as assessed by anti-Müllerian hormone (AMH)
Quality of life of cancer patients | up to one year
  Assessed by European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30(EORTC QLQ-C30)
Cancer specific rehabilitation | up to one year
  Assessed by Cancer rehabilitation evaluation system-short form (CARES-SF)
Reproductive concerns after cancer | up to one year
  Assessed by Reproductive Concerns After Cancer (RCAC) scale. The minimum and maximum values are 18 and 90 respectively, and a higher score means a higher level of reproductive concern or anxiety

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No